CLINICAL TRIAL: NCT03327467
Title: Expanded Access Protocol: Umbilical Cord Blood Infusions for Children With Brain Injuries
Status: Available | Type: Expanded Access
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00083888
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy; Hydrocephalus; Apraxia of Speech; Hypoxia Ischemia, Cerebral; Drowning; Anoxia
MeSH Terms: conditions — Cerebral Palsy; Hydrocephalus; Apraxias; Hypoxia-Ischemia, Brain; Drowning; Hypoxia

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Cord Blood Infusion — IV infusion of umbilical cord infusion (sibling, autologous, or unrelated donor)

SUMMARY:
This protocol is designed to enable access to intravenous infusions of banked umbilical cord blood (CB), that is thawed and not more than minimally manipulated, for children with various brain disorders. Children with cerebral palsy, congenital hydrocephalus, apraxia, stroke, hypoxic brain injury and related conditions will be eligible if they have normal immune function and do not qualify for, have previously participated in, or are unable to participate in an active cell therapy clinical trial at Duke Medicine. For the purpose of this protocol the term children refers to patients less than 26 years of age. Cord blood is administered as a cellular infusion without prior treatment with chemotherapy or immunosuppression. The mechanism of action is through paracrine signaling of cord blood monocytes inducing endogenous cells to repair existing damage.

DETAILED DESCRIPTION:
The primary purpose of this protocol is to enable access to autologous (a person's own) or allogeneic (someone else's) umbilical cord blood infusion for children with various brain disorders. Children with cerebral palsy, hydrocephalus, hypoxic brain injury, stroke, apraxia, and other brain injuries may be eligible if they do not qualify for or are unable to participate in another active clinical trial at Duke. For the purpose of this protocol the term children refers to patients less than 26 years of age. Cord blood infusions are still being studied to determine if they are effective in helping to treat certain types of brain injuries.

If being seen at Duke, the participant will be enrolled on the screening protocol, "A Research Database and Screening Protocol for Children with Brain Injuries Potentially Undergoing Cellular Therapy or Other Clinical Trials". Information about the participant's health and eligibility will be obtained under this protocol and may include records such as diagnostic information, genetic testing, videos, pictures of the child, and a cord blood report. The study team will review these records to determine if the child and the cord blood unit are eligible. For all cord blood infusions, the unit must meet certain cell count, sterility, and viability criteria. For sibling and unrelated donor cord blood infusions, the intended recipient and their sibling must be at least a half HLA match, and in the case of an unrelated donor, a 4/6 match.

If eligible, the participant will come to the hospital with a parent or legal guardian for clinical evaluations and infusion of the umbilical cord blood unit. Typically, medical evaluations are done on day one of the visit and the infusion is given on day two. On the day of infusion, CB cells will be thawed and transported to the Pediatric clinic for infusion to the participant under the supervision of the treatment team and/or clinic staff. A peripheral IV will be placed. Some children may require numbing cream and/or intranasal or oral versed prior to IV placement. Prior to the infusion of cells, premedications (Benadryl, Solumedrol) will be administered. The CB will be infused over approximately 5-15 minutes using standard practices. The participant will receive maintenance IV fluids and be observed in the clinic for a minimum of thirty minutes after the infusion. Participants will be discharged from clinic after at least thirty minutes, providing all vital signs are at their baseline and they are awake, taking oral fluids, and asymptomatic with no evidence of toxicity.

If a participant has evidence of illness on the day of planned infusion, including but not limited to fever, vomiting, diarrhea, or respiratory distress, the infusion will be postponed.

In the event that a participant develops signs or symptoms of anaphylaxis including rash, difficulty breathing, cough, wheezing, or vomiting during their CB infusion, the infusion will be terminated or slowed and appropriate medical therapy initiated.

Parents will be required to participate in remote follow-up phone calls and be willing to complete questionnaires for safety follow ups. Safety questionnaires will be sent by email at one and two years after the infusion.

Required Evaluations:

1. Screening:

   1. blood counts, blood chemistries, participant HLA typing, blood type (for females receiving allogeneic CB units)
   2. confirmatory HLA typing of the cord blood unit
2. Baseline Visit:

   1. History and Physical Exam
   2. Pregnancy test (blood test for menstruating females)
   3. blood counts, blood chemistries, if not performed during screening or within 12 months prior to the baseline visit
   4. infectious disease testing, blood type, test for antibodies against donor blood type (for those receiving allogenic cord blood)
3. Safety Assessments

   1. phone call the day after the infusion
   2. email safety survey at 1 and 2 years after the infusion

Multiple CB infusions may be administered from the same or two unique CB donors, but subsequent infusions will depend upon the quality and availability of an autologous or sibling cord blood unit and the need to limit exposure of the participant to new HLA antigens.

1. Donor source(s):

   A participant may receive an infusion from a maximum of two non-self donors in the following combinations:
   * Two sibling donors
   * One sibling and one unrelated donor (in any sequence)

   If a participant receives an infusion from a second non-self donor, the second sibling or unrelated donor must be a full 6/6 HLA match with either the recipient and/or the first non-self donor.

   Two unique unrelated donors is NOT permissible.
2. Each cord blood unit used for infusion must meet the cord blood and donor screening criteria.
3. A single cord blood unit may be used for multiple sequential infusions if there are enough cells available.

ELIGIBILITY:
Under this protocol, participants may be eligible for infusion of autologous, sibling, and/or unrelated donor CB cells (Duke only). Some eligibility criteria vary based on CB source. For all participants, eligibility is predicated on the availability of a qualifying CB unit To be eligible, patients must:

Inclusion Criteria:

1. Age at Consent:

   1. Autologous: 0-26 years
   2. Sibling: 6 months - 26 years
   3. Unrelated Donor (Duke only): 6 months - 26 years
2. Diagnosis

   1. Autologous and Sibling: Cerebral palsy, Hypoxic brain injury, Stroke, Hydrocephalus, Apraxia (without autism), Other brain injury
   2. Unrelated Donor (Duke only): Motor impairment secondary to: Hypoxic brain injury, Periventricular leukomalacia, Stroke/bleed, Congenital hydrocephalus
3. Functional Status:

   1. Autologous and Sibling: See exclusion criteria
   2. Unrelated Donor (Duke only): GMFCS level I-IV (age ≥2)
4. No clinically significant abnormalities in blood counts and basic chemistries for age.
5. Absolute Lymphocyte Count:

   * 1200 for African American participants
   * 1500 for all other participants
6. Availability of a qualified autologous or Sibling CB Unit

   1. Autologous or Sibling: available
   2. Unrelated Donor (Duke only): N/A
7. Written informed consent obtained from the parent or legal guardian.

Exclusion Criteria:

1. Documented HIV or Hepatitis or other disease transmittable through the blood.
2. A cord blood unit that fails to meet specifications
3. Refusal of consent
4. Uncontrolled seizure disorder
5. Uncontrolled infection
6. Diagnosed with a genetic or metabolic disorder related to the neurologic condition
7. History of an immune deficiency
8. History of treatment with chemo or immunosuppressive therapy
9. History of previous allogeneic cell therapy outside of participation in a Duke clinical trial
10. Need for mechanical ventilation or chronic O2 support
11. Unstable airway
12. Eligible for an active clinical trial of cellular therapy at Duke. If previously enrolled on another Duke cell therapy protocol the participant may still be considered for enrollment on this study after the follow-up period for the clinical trial is completed.
13. Cerebral palsy secondary to infection, congenital or otherwise, without another known cause
14. Pregnant or breastfeeding
15. Treated with autologous cellular therapy through a non-intravenous route (ie. intrathecally) within one year prior to enrollment.

Umbilical Cord Blood Criteria

Participant enrollment is dependent on the availability of a banked unit of autologous or sibling CB that has been stored at a private or public bank, or, if enrolling at Duke, availability of a publicly banked unrelated donor unit. Units must meet the following criteria:

Precryopreservation:

1. TNCC ≥2x107/kg
2. Sterility cultures performed and negative
3. Viability ≥70%
4. At least haploidentical HLA match for sibling units and at least a 4/6 HLA match for unrelated donor units
5. Donor screening testing performed and negative

CBU Test sample

1. Segment or test vial available
2. Identity confirmed via HLA typing of test sample and donor
3. Viability testing recommended, but not required

Max Age: 26 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, Principal Investigator — Duke University; Jessica Sun, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Rutgers Cancer Institutute, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina